CLINICAL TRIAL: NCT02099734
Title: Germ Cell Tumor and Testicular Tumor DNA Registry
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-016
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Germ Cell Tumor; Testicular Tumor
Keywords: 14-016
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Testicular Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood saliva

GROUPS / COHORTS (3):
- A: suspicion of germ cell tumor and/or a testicular mass: patients with testicular GCTs and non-GCT testicular tumors, extragonadal male GCTs, and female GCTs,
  Interventions: Behavioral: Questionnaires; Other: sample of blood or saliva
- B: family members of Group A: relatives of patients with GCTs or testicular tumors
  Interventions: Behavioral: Questionnaires; Other: sample of blood or saliva
- C: healthy controls unrelated to Group A or B: healthy controls who are unrelated to Groups A or B and do not have a personal history of cancer nor a family history of GCT or non-GCT testicular tumors
  Interventions: Behavioral: Questionnaires; Other: sample of blood or saliva

INTERVENTIONS:
Behavioral: Questionnaires
Other: sample of blood or saliva — A sample of blood or saliva will be obtained for DNA extraction. Approximately 2-4 tubes of blood will be collected or one tablespoon of saliva. If a participant has already provided a DNA sample for another MSKCC IRB approved protocol, they may not need to provide an additional sample.

SUMMARY:
This study is being done to create a registry to help us learn more about germ cell tumors (GCT) and other testicular tumors. The registry will include people with these tumors and also relatives and unrelated people without these tumors. This study will help us learn more about the prevention, diagnosis, treatment and outcome of these tumors. Studying relatives of patients and people unrelated to patients with GCT and other testicular tumors will help us understand why some people get these tumors and why some people don't.

ELIGIBILITY:
Inclusion Criteria:

Case Cohort

* Must be ≥ 18 years of age AND
* Must be an English-speaker AND
* Must have a diagnosis or suspicion of germ cell tumor and/or a testicular mass

Family Member Cohort

* Must be ≥ 18 years of age AND
* Must be an English-speaker AND
* Must be a blood relative of the proband. Family members of probands are eligible. These individuals need not have a diagnosis of GCT-TT, as they will be used for segregation analysis of suspected variants found in the proband.

Control Cohort

* Must be ≥ 18 years of age AND
* Must be an English-speaker AND
* Must not have a personal history of cancer, with the exception of non-melanoma skin cancer, AND
* Must not have a family history of germ cell tumor or testicular tumor AND
* Must not be a blood relative of controls enrolled in this study

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At MSKCC, the following outpatient clinics will be used to recruit GCT and testicular tumor cases and controls: Urology (Department of Surgery), Gynecologic Oncology (Department of Surgery) Clinical Genetics, Genitourinary Oncology (Department of Medicine), and Gynecologic Medical Oncology (Department of Medicine).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
creation of a Germ Cell Tumor and testicular tumor registry | 5 years
  We will collect clinical data including diagnosis date, pathology, family history, and risk factors in patients with GCT-TT.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Feldman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Cold Springs Harbor Laboratory (Specimen Analysis), Cold Spring Harbor, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/